CLINICAL TRIAL: NCT01938417
Title: Tobramycin Exposure From Active Calcium Sulfate Bone Graft Substitute
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Francoise Livio, MD, Médecin associé, University of Lausanne Hospitals
Other Study IDs: Tobramycin cast
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Orthopedic Operations
Keywords: tobramycin; bone graft substitute; pharmacokinetics; renal failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tobramycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adult patients treated with Osteoset® T (tobramycin sulfate): 10 g or 20 g of Osteoset® T
  Interventions: Drug: tobramycin

INTERVENTIONS:
Drug: tobramycin

SUMMARY:
This study aimed to assess the systemic absorption and disposition of tobramycin in patients treated with a tobramycin-laden bone graft substitute (Osteoset® T).

ELIGIBILITY:
Inclusion Criteria:

* Adult (> or =18 years old) patients
* Treatment with Osteoset® T

Exclusion Criteria:

* Intravenous tobramycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients treated with Osteoset® T in our orthopedic surgery department
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Measurement of systemic tobramycin concentration | within 10 days after surgery
  Develop a population pharmacokinetic model for tobramycin in patients treated with an active calcium sulfate bone substitute and to predict tobramycin systemic exposure under various dose and renal function levels.

REFERENCES:
- [Derived] Livio F, Wahl P, Csajka C, Gautier E, Buclin T. Tobramycin exposure from active calcium sulfate bone graft substitute. BMC Pharmacol Toxicol. 2014 Mar 4;15:12. doi: 10.1186/2050-6511-15-12. PMID 24593819